CLINICAL TRIAL: NCT04583384
Title: Evolution of Succinate Accumulation Detected in Vivo by Spectroscopic Magnetic Resonance Imaging (1H-SRM) After External Beam Radiation Therapy in SDHx-mutated Patients With Cervical Paragangliomas
Brief Title: In Vivo Succinate Detection After External Beam Radiation Therapy in SDHx- Paragangliomas
Acronym: RADIOSUCCES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Society for Endocrinology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP200281; 2020-A00397-32 (Other: IDRCB)
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Paraganglioma of Head and Neck
Keywords: Paraganglioma,SDHx genes, 1H-Spectroscopy MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Intervention (Other): Addition to the cervical angio-MRI, of a sequence of 1H-SRM 3T (SUCCESS) centered on the lesion studied, performed according to the following parameters: PRESS asymmetric monovoxel "PROBE", TE 144 ms, TR 2500 ms, 768 or 1024 medium.
  Interventions: Diagnostic Test: 1H-Spectroscopy MRI

INTERVENTIONS:
Diagnostic Test: 1H-Spectroscopy MRI — PRESS asymetric monovoxel " PROBE ", TE 144 ms, TR 2500 ms, 768 or 1024 averages

SUMMARY:
Qualitative and quantitative biomarker of response to radiotherapy is needed in paragangliomas. We aim at assessing the added value of 1H-SRM for the evaluation of early response to EBR therapy in patients with cervical SDHx PGL.

DETAILED DESCRIPTION:
Paragangliomas (PGL) are rare neuroendocrine tumors inherited in 40% of cases. SDHx genes (SDHA, SDHB, SDHC, SDHD), encoding the 4 subunits of the mitochondrial enzyme succinate dehydrogenase (SDH), are the most frequently involved.

Accumulation of succinate, the substrate for SDH, is a very specific biomarker for these mutations. Recently, we have demonstrated the feasability of detecting and quantifying succinate in tumors in vivo, by magnetic resonance spectroscopy (1H-SRM).

Patients carrying these mutations frequently develop cervical PGL for which the treatment of choice is external beam radiation therapy (EBR).

The objective of this project is to determine the feasibility of using 1H-SRM for the evaluation of early response to EBR therapy in patients with cervical SDHx PGL.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed informed consent
* Patient with cervical PGL with planning of treatment with EBR
* Patient with an SDHx mutation or unknown genetic status
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Pregnant woman
* Contraindication to MRI (implantable device, etc.)
* Impossibility of lying down without movement for 45 minutes (hyperalgesic patient, claustrophobia, etc.)
* PPGL having previously been the subject of local (excluding surgery) or systemic treatment
* PPGL <1 cm longest axis
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Disappearance of succinate accumulation at M12 | 12 months
  Absence of succinate accumulation detected in vivo by 1H-SRM, in cervical PGLs with SDHx mutations, at 12 months after EBR, reviewed by 2 independant experts blinded to all other clinical and genetics data.

SECONDARY OUTCOMES:
Disapperance of succinate accumulation at M3 | 3 months
  Absence of succinate accumulation detected in vivo by 1H-SRM, in cervical PGLs with SDHx mutations, at 3 months after EBR, reviewed by 2 independant experts blinded to all other clinical and genetics data.
Performance of cervical MRI at M3 and M12 after EBR | 12 months
  Reference diagnostic for response assessed by MRI at 3 months and 12 months after EBR: 1/ Complete response : tumour disappearance ; 2/ Partial response : decrease by at least 30% of tumour volume and no clinical symptomatology worsening ; 3/ stable : stability of tumour size and no clinical symptomatology worsening; 4/ Progression : increase by at least 20% of tumour volume and/or clinical symptomatological worsening
Performance of PET/CT at M12 after EBR | 12 months
  PERCIST criteria (PET response criteria in solid tumors) assessed by PET/CT at 3 months and 12 months after EBR
Metastatic evolution or death at M12 | 12 months
  Occurence of an event related to the disease during 12 months follow-up (metastatic evolution of the disease or death). Metastases diagnostic is assessed remotely by presence in chromaffin tissue (http://www.sfendocrino.org/article/599/recommandations)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence AMAR, PhD, Principal Investigator — Hôpital Européen Georges-Pompidou
Locations (3):
- France (3):
  - Hôpital Lariboisière, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hopital européen Georges Pompidou, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization